CLINICAL TRIAL: NCT05284968
Title: Clinical Study on the Safety and Efficacy of RD07 Cell Injection in the Treatment of Patients With Advanced Claudin18.2 Positive Solid Tumors
Brief Title: RD07 Cell Injection in the Treatment of Patients With Advanced Claudin18.2 Positive Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD07-07
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; CAR-T
MeSH Terms: interventions — Carboxylesterase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cell injection (Experimental): Cell injection
  Interventions: Drug: Cell injection

INTERVENTIONS:
Drug: Cell injection — All subjects will be treated with cell injection

SUMMARY:
IP: RD07 cell injection; Target disease：solid tumor; Protocol design： Single arm, open label, dose increasing design. The experiment was divided into two stages: dose increasing stage and dose extension stage. After the completion of the dose escalation phase (9 or 12 cases) and the conclusion of safety, the investigator can select the appropriate dose group according to the safety, tolerance, and treatment response to enter the dose expansion phase. Dose extension stage (24 and 27 cases) according to the indications in the crowd into three queues: respectively for the integration of a stomach and the stomach esophagus adenocarcinoma, pancreatic cancer and other solid tumor, expand stage each queue number of cases can be determined by the actual filter and into the group of patients, no separate regulation, but two phase of the total case must not exceed 36 cases.

DETAILED DESCRIPTION:
Principle of dose escalation:

1. If there is no DLT in 3 subjects in one dose group, increase to the next dose group;
2. If DLT occurs in only 1 of 3 subjects in a dose group, 3 subjects will be added to the dose group. If no more than 1 out of 6 subjects developed DLT, then increments to the next dose group;
3. If DLT occurs in ≥2 of 6 subjects, the level of the dose group exceeds MTD and should be reduced to the first dose group. If there were only 3 patients in the dose group, 3 more patients were enrolled. If this dose has been tested in 6 patients, the test is over and this dose is MTD;
4. If the dose increase to the highest dose group still does not reach MTD, the dose increase should be stopped.

Dose extension After the completion of the dose escalation phase (9 or 12 cases) and the conclusion of safety, the investigator can select the appropriate dose group according to the safety, tolerance, and treatment response to enter the dose expansion phase. Dose extension stage (24 and 27 cases) according to the indications in the crowd into three queues: respectively for the integration of a stomach and the stomach esophagus adenocarcinoma, pancreatic cancer and other solid tumor, expand stage each queue number of cases can be determined by the actual filter and into the group of patients, no separate regulation, but two phase of the total case must not exceed 36 cases.

Multiple infusion Efficacy was assessed as PR or SD lasting more than 12 weeks after the initial infusion, and subsequent infusion could be considered if patients developed disease progression. The pretreatment plan before the second infusion is the same as the first pretreatment. The researcher can decide whether to preprocess and adjust the pretreatment plan according to the specific situation of the subjects. Re-infusion can be performed 48 hours after the completion of the re-infusion, and the follow-up nodes after the re-infusion are the same as the treatment cycle of the first infusion. If the efficacy evaluation of the subjects is still PD after the re-infusion, RD07 infusion will not be performed later.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18 years old and <75 years old, gender is not limited; 2) Claudin18.2 positive confirmed by histology or cytology (the proportion of positive cells is ≥10% and the staining intensity is ≥1+; the specimen is acceptable within 1 year, and re-biopsy is required for more than 1 year) advanced gastric cancer, gastroesophageal combination solid tumors such as adenocarcinoma and pancreatic cancer; 3) Patients with gastric cancer and gastroesophageal junction adenocarcinoma who are ineffective in second-line standard therapy, or who are unwilling to perform or cannot tolerate second-line standard therapy; pancreatic cancer patients who fail or cannot tolerate first-line therapy; for other tumor types patients, they should meet the requirements of the existing standard of care for ineffective or intolerable standard treatment; 4) Referring to the RECIST 1.1 standard, there is at least one measurable lesion: according to CT or MRI evaluation, the longest diameter of the lesion is at least 10 mm (slice thickness 5 mm); or the short diameter of the lymph node lesion must be ≥15 mm; 5) ECOG score 0-2 points; 6) Blood routine neutrophil count ≥1.5×109/L; hemoglobin ≥80g/L and platelets ≥75×109/L (no blood transfusion within 14 days); 7) Creatinine clearance rate > 60ml/min (Cockcroft and Gault formula); for patients without liver involvement, serum total bilirubin is less than or equal to 1.5 times the upper limit of the normal value, and both serum ALT and AST are less than or equal to 3 times the upper limit of the normal value range; For liver violations, serum total bilirubin is ≤3 times the upper limit of the normal value, and both serum ALT and AST are ≤5 times the upper limit of the normal value range; 8) Echocardiography shows left ventricular ejection fraction (LVEF) ≥ 50%; 9) The estimated survival period is more than 3 months; The subjects or their legal guardians voluntarily participated in this trial and signed the informed consent.

Exclusion Criteria:

* 1) Those who have received Claudin18.2-targeted monoclonal antibody or cell therapy in the past; 2) Uncontrolled intracranial metastases (except those with stable disease for ≥8 weeks and no need for glucocorticoid therapy within 4 weeks after the first dose); 3) Acute pancreatitis or severe active upper gastrointestinal disease history within 4 weeks, such as upper gastrointestinal bleeding, etc.; 4) Receive anti-tumor therapy before infusion, if any of the following are met, it should be excluded: Received chemotherapy and small molecule targeted therapy within 2 weeks; Received radiotherapy within 4 weeks; Have received monoclonal antibody treatment and the last monoclonal antibody infusion is less than 2 half-lives from apheresis;

  * Received traditional Chinese medicine, Chinese patent medicine, etc. for the main purpose of anti-tumor treatment within 1 week.

    5) Those who used granule/granule-monoline colony-stimulating factor (G/GM-GSF) within 2 weeks before screening; 6) Patients who must use steroid hormones during CAR-T infusion (except for topical or inhaled steroid hormones); patients who are receiving systemic steroid therapy before screening and who are judged by the investigator to need long-term use of systemic steroid therapy during treatment. subjects (except inhalation or topical use); and subjects treated with systemic steroids within 72 hours before cell infusion (except inhalation or topical use); 7) Those with a history of serious heart disease, including but not limited to: history of acute myocardial infarction within 12 months, unstable angina pectoris, chronic heart failure of grade ≥III (standard of New York Heart Association), and electrocardiogram showing QT History of prolonged interval or severe arrhythmia; 8) Those with a history of craniocerebral trauma, disturbance of consciousness, epilepsy, cerebrovascular ischemia, cerebrovascular hemorrhagic disease, etc.; 9) Uncontrolled severe active infection (except for simple urinary tract infection and bacterial pharyngitis); 10) Subjects with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood HBV DNA >1000 copies/ml at screening; hepatitis C virus (HCV) antibody positive or peripheral blood HCV RNA positive ; Human immunodeficiency virus (HIV) antibody positive; Syphilis antibody positive; 11) Autoimmune disease subjects in need of treatment or subjects in need of immunosuppressive treatment; 12) The subject has a history of other primary cancers, except for the following: Non-melanoma cured by resection, such as skin basal cell carcinoma; Cervical carcinoma in situ, local prostate cancer, and ductal carcinoma in situ with a disease-free survival period of ≥2 years after adequate treatment; 13) The subject has a history of alcoholism, drug addiction or mental illness; 14) Inoculated with live or attenuated or inactivated vaccine within 4 weeks before screening; 15) Those who have a history of allergy to any component in the cell product; 16) Those who have participated in other clinical trials within 2 weeks before screening; 17) Pregnant, lactating women and subjects who are fertile and cannot take effective contraceptive measures (whether male or female); Any other condition that the investigator believes may increase the risk to the subject or interfere with the results of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) | 3 years
Adverse events (TEAEs) and incidence after initial infusion, treatment-related adverse events and incidence, AESI and incidence of special concern | 3 years

SECONDARY OUTCOMES:
ORR | 3 years